CLINICAL TRIAL: NCT04072445
Title: Phase II Trial of Trifluridine/Tipiracil in Combination With Irinotecan in Biliary Tract Cancers
Brief Title: Trifluridine/Tipiracil and Irinotecan for the Treatment of Advanced Refractory Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1941; NCI-2019-05653 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1941 (Other: Mayo Clinic)
Record Dates: First submitted 2019-08-27; First posted 2019-08-28 (Actual); Results first posted 2022-09-22 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-07

CONDITIONS: Advanced Bile Duct Carcinoma; Advanced Gallbladder Carcinoma; Refractory Bile Duct Carcinoma; Refractory Gallbladder Carcinoma; Stage III Distal Bile Duct Cancer AJCC v8; Stage III Gallbladder Cancer AJCC v8; Stage III Intrahepatic Bile Duct Cancer AJCC v8; Stage IIIA Distal Bile Duct Cancer AJCC v8; Stage IIIA Gallbladder Cancer AJCC v8; Stage IIIA Intrahepatic Bile Duct Cancer AJCC v8; Stage IIIB Distal Bile Duct Cancer AJCC v8; Stage IIIB Gallbladder Cancer AJCC v8; Stage IIIB Intrahepatic Bile Duct Cancer AJCC v8; Stage IV Distal Bile Duct Cancer AJCC v8; Stage IV Gallbladder Cancer AJCC v8; Stage IV Intrahepatic Bile Duct Cancer AJCC v8; Stage IVA Gallbladder Cancer AJCC v8; Stage IVB Gallbladder Cancer AJCC v8
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Irinotecan; Trifluridine; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (trifluridine and tipiracil, irinotecan) (Experimental): Patients receive trifluridine and tipiracil hydrochloride PO BID on days 1-5 and irinotecan hydrochloride IV over 90 minutes on day 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Irinotecan; Drug: Irinotecan Hydrochloride; Drug: Trifluridine and Tipiracil Hydrochloride

INTERVENTIONS:
Drug: Irinotecan — Given IV
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U-101440E
Drug: Trifluridine and Tipiracil Hydrochloride — Given PO
  Other Names: Lonsurf; TAS 102; TAS-102; Tipiracil Hydrochloride Mixture with Trifluridine; Trifluridine/Tipiracil; Trifluridine/Tipiracil Hydrochloride Combination Agent TAS-102

SUMMARY:
This phase II trial studies how well trifluridine/tipiracil and irinotecan work in treating patients with biliary tract cancer that has spread to other places in the body (advanced) and has not responded to treatment (refractory). Trifluridine/tipiracil and irinotecan may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the efficacy of trifluridine and tipiracil hydrochloride (trifluridine/tipiracil) in combination with irinotecan hydrochloride (irinotecan) in patients with refractory biliary tract cancers using progression-free survival (PFS) at 16 weeks.

SECONDARY OBJECTIVES:

I. Assess the safety and tolerability of trifluridine/tipiracil in combination with irinotecan in patients with refractory biliary tract cancers through adverse event monitoring.

II. Further explore the efficacy of trifluridine/tipiracil in combination with irinotecan in patients with refractory biliary tract cancers by overall response rates (ORR), disease control rates (DCR), and overall survival (OS).

CORRELATIVE RESEARCH:

I. To determine if the number of circulating tumor cells (CTCs) or the level of cell-free deoxyribonucleic acid (DNA) (cfDNA) at baseline is prognostic or predictive to the response to therapy.

II. To determine if changes in CTCs or cfDNA correlate with efficacy endpoints. III. To determine if drug response from a parallel ex vivo trial using patient-derived tumor organoid correlates with clinical response to trifluridine/tipiracil plus irinotecan.

IV. To evaluate the role of thymidine kinase 1 (TK1) in predicting the clinical benefit of trifluridine/tipiracil plus irinotecan and discover potential mechanisms of resistance using patient-derived tumor organoid and pre-treatment biopsy specimen.

EXPLORATORY RESEARCH:

I. To evaluate patients who received prior treatment with fluorouracil (5-FU) independently from the entire population in the following areas: PFS, safety and tolerability, ORR, DCR, and OS.

OUTLINE:

Patients receive trifluridine and tipiracil hydrochloride orally (PO) twice daily (BID) on days 1-5 and irinotecan hydrochloride (IV) over 90 minutes on day 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 3 months for up to 2 years after study registration.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of advanced biliary tract cancers including cancers originating in the gallbladder who have received at least one line of systemic anticancer therapy

  * Note: Patients who have either progressed on or are intolerant to the prior therapy can be included in this study
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria

  * NOTE: Tumor lesions in a previously irradiated area are not considered measurable disease. Disease that is measurable by physical examination only is not eligible
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Absolute neutrophil count (ANC) >= 1500/mm^3 (=< 21 days prior to registration)
* Platelet count >= 100,000/mm^3 (=< 21 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (=< 21 days prior to registration)
* Aspartate transaminase (AST) or alanine transaminase (ALT) =< 3 x ULN (=< 21 days prior to registration)
* Creatinine =< 1.5 x ULN (=< 21 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willingness to provide mandatory blood and tissue specimens for correlative research

Exclusion Criteria:

* Any of the following because this study involves an agent that has potential genotoxic, mutagenic and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception for at least 3 months after the last dose of the study drug
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm =< 21 days prior to registration
* Receiving any anticancer therapy for biliary tract cancer =< 21 days prior to registration
* Other active malignancy requiring treatment in =< 6 months prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix
  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* History of myocardial infarction =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Previous treatment with irinotecan or irinotecan-based chemotherapy for biliary tract cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Mahipal, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Tella SH, Foster N, Qian S, Nguyen T, Borad MJ, McWilliams RR, Alberts SR, Wee Ma W, Chakrabarti S, Fruth B, Wessling J, Hartgers M, Washburn L, Fernandez-Zapico ME, Hogenson TL, Pitot H, Jin Z, Mahipal A. Phase II Trial of Trifluridine/Tipiracil Plus Irinotecan in Patients with Advanced, Refractory Biliary Tract Carcinoma. Oncologist. 2023 Oct 3;28(10):917-e966. doi: 10.1093/oncolo/oyad144. PMID 37339254
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Trifluridine and Tipiracil, Irinotecan): Patients receive trifluridine and tipiracil hydrochloride PO BID on days 1-5 and irinotecan hydrochloride IV over 90 minutes on day 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.>
  > Irinotecan: Given IV>
  > Irinotecan Hydrochloride: Given IV>
  > Trifluridine and Tipiracil Hydrochloride: Given PO
Period: Overall Study
Arm/Group | Treatment (Trifluridine and Tipiracil, Irinotecan)
Started | 28
Completed | 27
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Trifluridine and Tipiracil, Irinotecan)
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (9.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Prior treatment [Count of Participants; unit: Participants]
  1 | 10
  2 | 11
  3+ | 7
Primary Site of Tumor [Count of Participants; unit: Participants]
  Extrahepatic biliary tract cancer | 9
  Gallbladder | 3
  Intrahepatic | 16
Degree of differentiation [Count of Participants; unit: Participants]
  Moderately | 18
  Poorly differentiated | 10
ECOG Performance Status (PS) [Count of Participants; unit: Participants] — ECOG = 0: Fully active, able to carry on all pre-disease performance without restriction.
  ECOG = 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  ECOG = 0 is better. ECOG = 1 is worse.
  Participants
    0 | 4
    1 | 24
Prior treatment with fluoropyrimidine based regimen [Count of Participants; unit: Participants]
  Yes | 3
  No | 25
Metastatic Sites [Count of Participants; unit: Participants]
  Bone | 1
  Liver | 25
  Peritoneum | 3
  Lung | 4
  Nodal | 3
  Abdominal Wall | 1
  Interaortocaval LN | 2
  Pancreas | 1
  Perisplenic and Perihepatic | 1
  Soft tissue, adrenal gland. | 1
  abdominal wall, mesenteric node. | 1
  hepatic duct | 1
MedDRA disease code [Count of Participants; unit: Participants]
  Cholangiocarcinoma, intrahepatic and extrahepatic bile ducts (adenocarcinoma) | 24
  Gall Bladder Carcinoma | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Will be defined as the proportion of evaluable patients who are progression-free (stable disease, partial response, complete response) at 16 weeks and assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. Confidence intervals for the true success proportion will be calculated according to the approach of Clopper and Pearson.
Time Frame: Up to 16 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment (Trifluridine and Tipiracil, Irinotecan): Patients receive trifluridine and tipiracil hydrochloride PO BID on days 1-5 and irinotecan hydrochloride IV over 90 minutes on day 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  >
  > Irinotecan: Given IV
  >
  > Irinotecan Hydrochloride: Given IV
  >
  > Trifluridine and Tipiracil Hydrochloride: Given PO
Arm/Group | Treatment (Trifluridine and Tipiracil, Irinotecan)
Number analyzed (Participants) | 27
percentage of participants | 37.0 [19.4 to 57.6]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Will be defined as the proportion of patients who experience either a partial response or complete response as their best response. ORR will be reported descriptively and a 95% confidence interval will be reported.
Time Frame: Up to 20 months
Population: 7 patients went off treatment early on and weren't evaluated for response post-baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Trifluridine and Tipiracil, Irinotecan)
Number analyzed (Participants) | 20
percentage of participants | 20.0 [5.7 to 43.7]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Will be defined as the proportion of patients who experience a partial response, complete response, or have stable disease as their best response. DCR will be reported descriptively and a 95% confidence interval will be reported.
Time Frame: Up to 20 months
Population: 7 patients went off treatment early on and weren't evaluated for response post-baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Trifluridine and Tipiracil, Irinotecan)
Number analyzed (Participants) | 20
percentage of participants | 50 [27.2 to 72.8]

4. Secondary Outcome: PFS
Description: Will be determined based on RECIST v 1.1. PFS will be estimated using the Kaplan-Meier method. The median PFS and 95% confidence interval will be reported. Patients will be censored at the last disease assessment date.
Time Frame: From study entry to the first of either disease progression or death from any cause, assessed up to 20 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Trifluridine and Tipiracil, Irinotecan)
Number analyzed (Participants) | 27
months | 3.9 [2.5 to 7.4]

5. Secondary Outcome: Overall Survival (OS)
Description: Will be estimated using the Kaplan-Meier method. The median OS and 95% confidence interval will be reported. Patients will be censored at the date patient was last known to be alive.
Time Frame: From study entry to death from any cause, assessed up to 20 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Trifluridine and Tipiracil, Irinotecan)
Number analyzed (Participants) | 27
months | 9.1 [8.0 to 14.3]

6. Secondary Outcome: Number of Participants With Adverse Events
Description: The maximum grade for each type of adverse event by patient will be summarized by frequencies and percentages using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Trifluridine and Tipiracil, Irinotecan)
Number analyzed (Participants) | 27
Participants
  Grade 3+ AE | 20
  Grade 4 AE | 4
  Grade 5 AE | 0

7. Other Pre Specified Outcome: Circulating Tumor Cells (CTCs) or Cell-free Deoxyribonucleic Acid (cfDNA) at Baseline
Description: Will determine if CTCs or cfDNA at baseline will correlate with prognosis or response to therapy.
Time Frame: Baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in CTCs or cfDNA
Description: Will determine if change in CTCs or cfDNA will correlate with efficacy endpoints.
Time Frame: Baseline up to 20 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Correlation of Response
Description: Will determine if drug response from a parallel ex vivo trial using patient-derived tumor organoid correlates with clinical response to trifluridine and tipiracil hydrochloride (trifluridine/tipiracil) plus irinotecan hydrochloride (irinotecan).
Time Frame: Up to 20 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Prediction of Clinical Benefit by Thymidine Kinase 1 (TK1)
Description: Will evaluate the role of TK1 in predicting the clinical benefit of trifluridine/tipiracil plus irinotecan and discover potential mechanisms of resistance using patient-derived tumor organoid and pre-treatment biopsy specimen.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 20 months
Arm/Group | Treatment (Trifluridine and Tipiracil, Irinotecan)
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 11/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Trifluridine and Tipiracil, Irinotecan) (N=27)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Ascites (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Biliary tract infection (Infections and infestations) | 3 (3)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Trifluridine and Tipiracil, Irinotecan) (N=27)
Anemia (Blood and lymphatic system disorders) | 26 (208)
Ascites (Gastrointestinal disorders) | 2 (6)
Diarrhea (Gastrointestinal disorders) | 6 (9)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 9 (19)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 4 (20)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Blood bilirubin increased (Investigations) | 2 (5)
Lymphocyte count decreased (Investigations) | 14 (59)
Neutrophil count decreased (Investigations) | 18 (34)
Platelet count decreased (Investigations) | 17 (90)
White blood cell decreased (Investigations) | 13 (29)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (5)
Dysgeusia (Nervous system disorders) | 3 (3)
Paresthesia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 4 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT04072445/Prot_SAP_000.pdf